CLINICAL TRIAL: NCT01149694
Title: A Randomized, Double-Blind, Parallel-Group, Single-Ascending Dose, Placebo-Controlled Safety and Tolerability Study of PUR 0110 Rectal Enema in Normal Healthy Volunteers
Brief Title: A Study to Assess the Safety and Tolerability of PUR 0110 Rectal Enema in Normal Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PurGenesis Technologies Inc. (Industry)
Responsible Party: André P. Boulet, PhD / President & Chief Operating Officer, PurGenesis Technologies, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PG08-PUR 0210-FIM001; 2009-010405-36 (EudraCT Number)
Record Dates: First submitted 2010-06-22; First posted 2010-06-23 (Estimated); Last update posted 2010-06-24 (Estimated); Status verified 2010-06

CONDITIONS: Ulcerative Colitis
Keywords: PurGenesis Technologies Inc.; PUR 0110 rectal enema; Ulcerative colitis; Distal; Normal healthy volunteers
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Other)
  Interventions: Drug: PUR 0110 Rectal Enema or Placebo Enema
- Cohort 2 (Other)
  Interventions: Drug: PUR 0110 Rectal Enema or Placebo Enema
- Cohort 3 (Other)
  Interventions: Drug: PUR 0110 Rectal Enema or Placebo Enema
- Cohort 4 (Other)
  Interventions: Drug: PUR 0110 Rectal Enema or Placebo Enema

INTERVENTIONS:
Drug: PUR 0110 Rectal Enema or Placebo Enema — 187.5 mg/60 g
  Other Names: PUR 0110 Enema; PUR 0110
  Arms: Cohort 1
Drug: PUR 0110 Rectal Enema or Placebo Enema — 375 mg/60 g
  Other Names: PUR 0110 Enema; PUR 0110
  Arms: Cohort 2
Drug: PUR 0110 Rectal Enema or Placebo Enema — 750 mg/60 g
  Other Names: PUR 0110 Enema; PUR 0110
  Arms: Cohort 3
Drug: PUR 0110 Rectal Enema or Placebo Enema — 1500 mg/60 g
  Other Names: PUR 0110 Enema; PUR 0110
  Arms: Cohort 4

SUMMARY:
This is a first-in-man study of a novel investigational botanical drug complex, PUR 0110 rectal enema, that has been shown to have potent anti-inflammatory, antioxidant and immunomodulatory effects following in vitro and in vivo pharmacology studies, to assess the safety and tolerability of sequential single-ascending doses in normal healthy volunteers and to determine the maximum tolerated dose (MTD). As a tertiary objective, the study will also investigate the presence of specific pharmacokinetic markers following the administration of single-dose PUR 0110 at each dose level.

The study is designed as a single-center, randomized, double-blind, parallel-group, sequential single-ascending dose, placebo-controlled safety, tolerability and pharmacokinetic study of PUR 0110 rectal enema in 24 normal healthy male volunteers. Eligible subjects will be randomly assigned to 4 Cohorts of 6 subjects each to receive active drug (PUR 0110 Enema) or placebo enema as follows: 187.5 mg/60 g - Cohort 1, 375 mg/60 g - Cohort 2, 750 mg/60 g - Cohort 3 or 1500 mg/60 g - Cohort 4. Within each Cohort, subjects will be randomized in a 2:1 ratio to receive either active treatment (PUR 0110 enema; n = 4) or placebo enema (n = 2). Each subject will receive only 1 dose of assigned study medication and dosing of subjects within each cohort will also be by sequential inclusion.

DETAILED DESCRIPTION:
Flexible sigmoidoscopy will be performed during the Screening Period within 72 to 48 hours pre-dose and within 9 +/- 1 hours post-dosing to visually examine the colonic mucosa for any signs of local toxicity and grade it as normal/abnormal; and 3 pinch biopsies will be obtained at each endoscopy at about the same level in the colon (<50 cm from the anal verge) for histology. At the baseline flexible sigmoidoscopy, subjects must have normal colonic and rectal mucosa (i.e., no bleeding, inflammation, edema, ulceration or other abnormal finding) to be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult non-smoking male volunteers between the ages of 18 to 55 years, inclusive.
* Must provide a voluntary written informed consent prior to initiation of screening, must be capable of following the verbal and written study instructions, and be able to commit to any confinements and return visits during the entire period of the study.
* Must have a body mass index (BMI) that is within 18 to 30 kg/m2 on the BMI Chart.
* Must have a normal digital rectal examination at screening.
* Must have normal colonic and rectal mucosa at the baseline flexible sigmoidoscopy (i.e., no bleeding, inflammation, edema, ulceration or other abnormal finding).
* Must have no clinically significant abnormal findings in their medical history, physical examination or clinical laboratory test results.

Exclusion Criteria:

* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatological, neurological, or psychiatric disease.
* History of allergic reaction or hypersensitivity to spinach, spinach tablet, spinach powder or spinach extract; and to latex, molds and mushrooms.
* Subjects with abnormal digital rectal examination at screening
* Subjects with abnormal colonic and rectal mucosa at the baseline flexible sigmoidoscopy i.e., have bleeding, inflammation, edema or ulceration or other abnormal finding.
* Subjects who used NSAIDs within 14 days prior to dosing.
* History of pseudoallergic hypersensitivity to the food color additives, tartrazine (E102) and sunset yellow (E110), allergic asthma, aspirin intolerance, and severe or multiple allergies.
* History of gout, pseudogout or hyperuricemia.
* History of kidney stones.
* Past medical history of significant colonic surgery, except for benign polyp removal.
* Subjects with anatomical abnormalities of the colon, e.g., short bowel or other abnormalities.
* Subjects with a history of rectal bleeding, passage of mucus rectally, and irregular bowel habits, e.g., frequent diarrhea or constipation.
* Subjects with internal or external hemorrhoids.
* History or presence of alcoholism or drug abuse within the past 2 years.
* Subjects with a current history of smoking. If a former smoker, must have stopped smoking for at least 3 months to qualify for study entry.
* Subjects who tested positive at screening for HIV, HbsAg or HCV.
* Subjects who used any prescription medications within 14 days prior to dosing.
* Subjects who used any rectal enema or laxative within 7 days prior to dosing.
* Subjects who used any over-the-counter (OTC) medications within 7 days prior to dosing.
* Subjects who have made a donation of blood or blood products (with the exception of plasma as noted below) within 56 days prior to dosing.
* Subjects who have made a plasma donation within 7 days prior to dosing.
* Subjects with hemoglobin less than 14.0 g/dl.
* Subjects who participated in another clinical trial within 28 days prior to dosing.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Incidence, nature and severity of adverse events and abnormal clinical laboratory test results | After single-ascending doses

SECONDARY OUTCOMES:
Maximum tolerated dose (MTD) | After single-ascending doses
Pharmacokinetic profile and parameters - if specific pharmacokinetic markers are successfully identified | After single-ascending doses

CONTACTS AND LOCATIONS:
Overall Officials: Theophilus J Gana, MD, PhD, Study Director — PurGenesis Technologies Inc.; Sergej Berger, MD, Principal Investigator — FOCUS Clinical Drug Development GmbH
Locations (1):
- FOCUS Clinical Drug Development GmbH Phase 1 Clinic, Neuss, Germany